CLINICAL TRIAL: NCT05218785
Title: Botulinum Toxin Injection As Treatment for Proximal Medial Gastrocnemius Muscle Tightness with Subsequent Chronic Plantar Fasciitis - a Prospective Clinical Cohort Study
Brief Title: Treatment of Gastrocnemius Tightness and Subsequent Chronic Plantar Fasciitis with Botulinum Toxin a
Acronym: PLATOX
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Ellingsen Husebye, MD PhD, Oslo University Hospital
Other Study IDs: REK351430
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Plantar Fascitis; Gastrocnemius Tightness
Keywords: proximal medial gastrocnemius recession; gastrocnemius tightness; botox; botulinum toxin a
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Botulinum toxin A injection: Patients will receive a total of 3 -three - injections of 75 IU Botulinum Toxin A in the proximal medial gastrocnemius muscle. Treatments will be performed by a specialist in neurology as a Ultra-Sound guided injection into the proximal medial gastrocnemius muscle Injections will be administered at baseline, 3 months and 6 months.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — 75 U in medial gastrocbemius head. x 3

SUMMARY:
This prospective clinical cohort study will follow 40 patients who recieve botulinum toxin A treatment for proximal medial gastrocnemius tightness with subsequent Chronic Plantar Fasciitis for two years. Three injections of botulinum toxin (75IU) will be administered with intervals of three months. Participants will be followed at baseline, 3 months, 6 months, 1 year and 2 years with Patient Related Outcome Measures (PROMS) and physical test (Ergotest and ankle dorsiflexion).

DETAILED DESCRIPTION:
The connection between gastrocnemius tightness and plantar fasciitis has been demonstrated in several clinical studies. Patients with chronic pathology, and unsatisfactory results from physical therapy, may benefit from gastrocnemius lengthening. This is usually obtained with proximal medial gastrocnemius recession surgery (PMGR), but recent studies and recent experience from our hospital suggest that similar effect may be obtained with ultrasound guided- injections of Botulinum Toxin A injections in the proximal medial gastrocnemius muscle.

This study will follow patients with gastrcnemius tightness (demonstrated by the Silferskiolds test) and subsequent chronic (MRI-verified) plantar fasciitits who has not recieved satisfactiory results from at least three months of guided physcial therapy.

Participants will recieve three ultrasound guided injections of 75IU of Botulinum Toxin A with three month intervals.

They will be followed with clinical controls for two years after the first injection.

THe main outcome is the Manchester Oxford Foot Questionnaire (MOxFQ).

ELIGIBILITY:
Inclusion criteria:

1. Age 18-75 years.
2. An isolated gastrocnemius contracture must be verified with the Silfverskiölds test before inclusion.
3. Diagnosis plantar fasciitis verified clinically by an orthopaedic surgeon.
4. Diagnosis verified by MRI. MRI criteria: Thickening of the plantar fascia, oedema in the calcaneus, pathological signal changes in the plantar fascia (35)
5. Duration of symptoms must be at least 12 months prior to first BTA injection.
6. Conventional Physical Therapy must have been tried at least three months without a significant reduction of symptoms in the affected foot.

Exclusion criteria:

1. Previously undergone surgery for plantar fasciitis.
2. Patients with severe talocrural pathology or serious malalignment of foot and ankle
3. Severely reduced peripheral circulation
4. History of alcoholism, drug abuse, psychological or other emotional problems likely to jeopardize informed consent.
5. Patients with a contraindication/non-compliance for MRI examination.
6. History of allergic reaction/anaphylactic reaction or other contraindication to botulinum toxin.
7. Not able to read and/or speak a Scandinavian language or English adequately.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of patients who recieve routine care at our hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Manchester Oxford Foot Questionnaire | 2 years
  MOxFQ (Manchester Oxford Foot Questionnaire) is a PROM consisting of 16 questions in three domains (pain, walking/standing, social interaction) leading to a total score from 0-100, 0 being the best possible score. It is validated as a reliable tool to measure results of foot and ankle surgery

SECONDARY OUTCOMES:
Achilles function test battery | 2 years
  The test battery consists of three jump tests, a counter movements jump (CMJ), a drop counter movement jump (drop CMJ) and hopping, and two strength tests, concentric toe-raises (resistance 13+23 kg), eccentric-concentric toe-raises (resistance 13+23 kg) and toe-raises for endurance. All recorded through the MuscleLab software.
Ankle dorsiflexion | 2 years
  measured by device that measures the ankle's range of motion that has been previously tested and found to be valid, reliable, and responsive in detecting isolated gastrocnemius contractures (IGCs). (40) An electric goniometer, Biometrics SG150 (Units 25-26, Biometrics Ltd, Newport, UK), with an accuracy of ±2 degrees and a repeatability of 1 degree will be used. The device will be calibrated before every new participant. Force applied directly beneath the head of the second metatarsal until the end range of dorsiflexion with a dynamometer.
Visual Analogue Scale (VAS) | 2 years
  Visual Analogue Scale for pain during use om affected leg in the last 24 hours. 0 is no pain. 10 is worst pain imaginable
EQ5D5L | 2 years
  Quality of life is measured by the EuroQol questionnaire (EQ-5D). EQ-5D is a validated generic health-related quality-of-life instrument. It consists of two parts: EQ-5D descriptive part and EQ-5D visual analogue scale. The descriptive part includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with three possible answers ("no problems", "some problems", and "major problems"). EQ5D VAS is a visual analogue scale of self-related overall health, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state)
AOFAS (American Orthopeadic Foot and Ancle Society) hindfoot score | 2 years
  AOFAS score measures pain, function, movement and deformity. It ranges from 0-100, 100 being the best possible score. The score is in our opinion not especially fit to measure the symptoms and change in symptoms in plantar fasciitis patients, but we include it to be able to compare our results to Abassain et al.
Adverse events | 2 years
  . I.e. infection, nerve injury, thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Orthopedic Department Ullevål, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No